CLINICAL TRIAL: NCT07160816
Title: A Real-world, Multi-centre, Prospective, Non-interventional, Single-arm Study Investigating Glycaemic Control, Treatment Satisfaction and Adherence Associated With the Use of Insulin Icodec in People Living With Type 1 Diabetes
Brief Title: A Research Study to See How Insulin Icodec Helps People With Type 1 Diabetes Control Their Blood Sugar
Status: Recruiting | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN1436-8404; U1111-1316-7988 (Other: World Health Organization (WHO))
Record Dates: First submitted 2025-08-29; First posted 2025-09-08 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — insulin icodec

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Insulin icodec: Participants with T1D will be treated with commercially available insulin icodec according to routine clinical practice at the discretion of the treating physician.
  Interventions: Drug: Insulin icodec

INTERVENTIONS:
Drug: Insulin icodec — Participants with T1D will be treated with commercially available insulin icodec.
  Other Names: Awiqli

SUMMARY:
The study will look at how well insulin icodec controls blood sugar levels in participants who have never used it before. Participants with type 1 diabetes (T1D) will be treated with insulin icodec as prescribed to by their doctor, in accordance with usual clinical practice. This study will last for about 22 to 30 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Signed consent obtained before any study-related activities (study-related activities are any procedures related to recording of data according to the protocol).
* The decision to initiate treatment with commercially available insulin icodec has been made by the participant/legally acceptable representative (LAR) and the treating physician before and independently from the decision to include the participant in this study.
* Male or female, age greater than or equal to (≥) 18 years at the time of signing informed consent.
* Diagnosed with T1D ≥ 1 year before signing informed consent.
* Treated with multiple daily insulin injections (daily basal insulin analogue and bolus insulin analogue regimen) ≥ 6 months before signing informed consent.
* Available HbA1c value less than or equal to (≤) 90 days prior to the 'Initiation visit' (V1) or HbA1c measurement taken in relation with the 'Initiation visit' (V1) if in line with local clinical practice.
* Treatment naïve to once-weekly insulin prior to the 'Initiation Visit' (V1).

Exclusion Criteria:

* Previous participation in this study. Participation is defined as having given informed consent in this study.
* Treatment with any investigational drug within 30 days prior to enrolment into the study.
* Mental incapacity, unwillingness or language barriers precluding adequate understanding or cooperation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population comprises participants who are diagnosed with type 1 diabetes and agree to be treated with insulin icodec after consultation with their physician independently from the decision to participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 245 (Estimated)
Dates: Start 2025-08-28 (Actual); Primary Completion 2027-01-20 (Estimated); Study Completion 2027-01-20 (Estimated)

PRIMARY OUTCOMES:
Change in glycated haemoglobin (HbA1c) | Baseline (week 0), week 26
  Measured as percentage (%) point of HbA1c.

SECONDARY OUTCOMES:
Change in Insulin Treatment Satisfaction Questionnaire (ITSQ) score | Baseline (week 0), end of study (week 22-30)
  ITSQ measures insulin treatment satisfaction, applicable to a wide range of insulin therapies. The ITSQ consists of 22 items yielding 5 domain scores and a total score. The domains consist of Regimen inconvenience (5 items), Lifestyle flexibility (3 items), Glycemic control (3 items), Hypoglycemic control (5 items), and Satisfaction with the insulin delivery device (6 items). The domain and global ITSQ score both ranges from 0-100.Higher scores indicate a better health state (less negative impact).
Change in Adelphi Adherence Questionnaire (ADAQ) score | Baseline (week 0), end of study (week 22-30)
  The ADAQ measure consists of 11 items scored on a scale of 0 to 4. The mean of the individual items represents the total ADAQ score. At least 8 of the 11 items must be answered to calculate the ADAQ score. The lower the score corresponds to the greater adherence.
Number of self-reported overall severe hypoglycaemia | From baseline (week 0) to end of study (week 22-30)
  Measured as number of episodes.
Clinical success as perceived by the physician | From baseline (week 0) to end of study (week 22-30)
  Measured as count of participant per response option.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (35):
- Germany (23):
  - Hausärztliche und Diabetologische Praxis Pirna, Pirna, LÄK Sachsen
  - Zuckerpraxis Dr. Ewald Jammers, Bramsche
  - Studiengesellschaft Dres. Könemann/Steinmann GbR, Bünde
  - Diabeteszentrum-Do Dres. K U. Ch. Busch GbR, Dortmund
  - Diabeteszentrum Duisburg-Mitte, Duisburg
  - MVZ im Altstadt-Carree Fulda GmbH - Zentrum für klinische Studien, Fulda
  - Gemeinschaftspraxis Dr. Martin Grüneberg, Herne
  - Mesut Durmaz, Hof, Hof
  - Dr. Carola Lüke, Jerichow
  - Diabetespraxis Kiel, Kiel
  - Praxis Am Oberen Tor - Dr. Simon-Wagner, Lichtenfels
  - Diabetologie Dr. Eidenmüller, Marburg
  - Dr. Bernhard Landers, Mayen
  - Diabeteszentrum Bogenhausen, München
  - Medicover Neu-Ulm MVZ, Neu-Ulm
  - Diabetespraxis Oranienburg, Oranienburg
  - Diabetesschwerpunktpraxis Dr. Martina Lange, Rheinbach
  - Med.Versorgungszentrum Riesa-Dr. Bieler, Riesa
  - Dr. med. Carsten Schürfeld, GZ-Vauban, Saarlouis
  - Diabetespraxis Schorndorf Dr. Hensel, Schorndorf
  - Praxis Dr. Zimmermann, Sonsbeck
  - Endokrinologikum Ulm, Ulm
  - Diabetespraxis Viersen, Viersen
- Italy (12):
  - Ospedale San Raffaele S.r.l. - Unità Clinica Endocrinologia, Milan, Lombardy
  - Azienda Sanitaria Locale Città di Torino - Ambulatorio Endocrinologia e Malattie Metaboliche, Turin, Piedmont
  - AUSL Toscana Nord Ovest - Ospedali Riuniti di Livorno - Diabetologia e Malattie del Metabolismo, Livorno, Tuscany
  - AUSL Toscana Nord Ovest - Cittadella della Salute Campo di Marte - Diabetologia Lucca e Valle del Serchio, Lucca, Tuscany
  - Azienda Ospedaliera Papa Giovanni XXIII, Bergamo
  - Azienda Ospedaliero-Universitaria Renato Dulbecco, Catanzaro
  - Azienda Ospedaliera Luigi Sacco, Milan
  - A.O.U. Università Studi della Campania "Luigi Vanvitelli", Naples
  - Azienda Ospedaliera di Perugia;Ospedale S. Maria della Misericordia, Perugia
  - DIABETOLOGIA Ravenna AUSL della Romagna, Ravenna
  - Universita Degli Studi Di Roma La Sapienza - Policlinico Umberto I Medicina Sperimentale, Roma
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS - Dipartimento di scienze Mediche e Chirurgiche, Rome

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: https://novonordisk-trials.com